CLINICAL TRIAL: NCT03114540
Title: A Phase 1, Open-Label Study to Characterize the Pharmacokinetics and Safety of a Single Oral Dose of GBT440 in Subjects With Hepatic Impairment
Brief Title: Single-Dose PK and Safety Study of GBT440 in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GBT440-0112; C5341047 (Other: Alias Study Number)
Record Dates: First submitted 2017-03-28; First posted 2017-04-14 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — voxelotor

STUDY DESIGN:
Intervention Model Description: Multiple-center, nonrandomized, open-label, parallel group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GBT440 Dose 1:Mild hepatic impairment (Experimental): Child Pugh A
  Interventions: Drug: GBT440
- GBT440 Dose 1:Moderate hep. impairment (Experimental): Child Pugh B
  Interventions: Drug: GBT440
- GBT440 Dose 1:Severe hepatic impairment (Experimental): Child Pugh C
  Interventions: Drug: GBT440
- GBT440 Dose 1:Normal hepatic function (Experimental): Healthy subjects
  Interventions: Drug: GBT440

INTERVENTIONS:
Drug: GBT440 — Oral

SUMMARY:
A Phase 1, multiple center, nonrandomized, open-label, parallel group study of a single oral dose of GBT440 administered in subjects with mild (Child-Pugh A), moderate (Child-Pugh B), or severe (Child-Pugh C) hepatic impairment disease and healthy subjects with normal hepatic function.

DETAILED DESCRIPTION:
Approximately 24 to 28 subjects will be enrolled. Safety and PK assessments will be performed at selected time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Males or females, 18 to 75 years old
* Willing and able to give written informed consent

Patients with hepatic impairment:

* Mild hepatic impairment (Child-Pugh A [5-6 points])
* Moderate hepatic impairment (Child-Pugh B [7-9 points])
* Severe hepatic impairment (Child-Pugh C [10-15 points])

Healthy subjects:

* Match in age, gender and body mass index with hepatic impaired subjects
* Healthy and without clinically significant abnormalities in vital signs, ECGs, physical exam, clinical laboratory evaluations, medical and surgical history

Exclusion Criteria:

All subjects:

* Participation in another clinical trial of an investigational drug (or medical device) within 30 days of the last dose of investigational drug or 5 half-lives whichever is longer, prior to screening, or is currently participating in another trial of an investigational drug (or medical device)
* Any signs or symptoms of acute illness at screening or Day -1
* History or presence of clinically significant allergic, hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease

Patients with hepatic impairment:

* History of liver transplantation, hepatic mass suggestive of hepatocellular carcinoma or acute liver disease
* Screening serum ALT or AST >5 times the upper limit of normal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
To assess the Cmax of GBT440 in patients with mild, moderate, or severe hepatic impairment | 28 days max
  Maximum observed plasma concentration
To assess the Tmax of GBT440 in patients with mild, moderate, or severe hepatic impairment | 28 days max
  Time at which maximum concentration was observed
To assess the AUC of GBT440 in patients with mild, moderate, or severe hepatic impairment | 28 days max
  Area under the concentration-time curve
To assess the T1/2 of GBT440 in patients with mild, moderate, or severe hepatic impairment | 28 days max
  Terminal elimination half-life

SECONDARY OUTCOMES:
Adverse events | 28 days max
Clinical laboratory tests | 28 days max
Physical examination findings | 28 days max
Vital signs | 28 days max
Electrocardiograms | 28 days max

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - OCRC, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-0112